CLINICAL TRIAL: NCT03022656
Title: A Randomized Clinical Trial of Brace Treatment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID Pandemic
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00058476
Record Dates: First submitted 2017-01-12; First posted 2017-01-16 (Estimated); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Scoliosis; Idiopathic, Infantile
Keywords: Orthotic treatment, Ultrasound Imaging
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monitor Only (Active Comparator): A brace monitor will be embedded inside the brace to monitor compliance.
  Interventions: Device: Active Brace system
- Active Brace System (Active Comparator): An active brace device will be embedded inside the brace to dynamically control interface pressure and monitor compliance.
  Interventions: Device: Active Brace system

INTERVENTIONS:
Device: Active Brace system

SUMMARY:
Brace treatment is the most effective non-surgical method for the treatment of Adolescent idiopathic scoliosis (AIS). The goal of bracing is to stop the curve progression during the high risk period of the adolescent growth spurt. A spinal brace is a hard plastic shell with pressure pads installed inside the liner to provide mechanical support to the curvature of the spine. It is a big commitment for adolescents to wear a brace because it is physically restrictive, uncomfortable and draws unwanted attention. Therefore, it is very important to make the brace treatment as effective as possible to get patient buy-in to compromise their lifestyle by wearing a brace. Patients' belief in the treatment outcomes is also a factor to attain their compliance.

This randomized clinical study will investigate if the effectiveness of brace treatment can be maximized by combining ultrasound imaging assistance during brace design with the smart brace to automatically maintain corrective brace pressures at the optimum level during the whole treatment period.

DETAILED DESCRIPTION:
Background: Brace treatment is the most effective non-surgical method for the treatment of AIS. The goal of bracing is to stop the curve progression during the high risk period of the adolescent growth spurt. A spinal brace is a hard plastic shell with pressure pads installed inside the liner to provide mechanical support to the curvature of the spine. It is a big commitment for adolescents to wear a brace because it is physically restrictive, uncomfortable and draws unwanted attention. Therefore, it is very important to make the brace treatment as effective as possible to get patient buy-in to compromise their lifestyle by wearing a brace. Patients' belief in the treatment outcomes is also a factor to attain their compliance.

Study Objective: This randomized clinical study will investigate if the effectiveness of brace treatment can be maximized by combining ultrasound imaging assistance during brace design with the smart brace to automatically maintain corrective brace pressures at the optimum level during the whole treatment period.

Methodology:

Subject Selection: One hundred and twenty-eight brace candidates with AIS will be recruited over the next 5 years. During the scoliosis clinic, the attending orthopaedic surgeon identifies a potential candidate. He will ask the potential patient if he/she is interested in speaking with the research coordinator about research projects that he/she is eligible. The inclusion criteria are patients 1) age 10 - 16 years, 2) diagnosis of AIS, 3) require full-time brace wear, 4) Cobb angle between 20° - 40°, 5) Risser sign ≤3 and 6) premenarchal or less than 1 year postmenarchal. Subjects will be randomly selected to 1 of the 2 groups: a) An ultrasound assisted designed brace and a brace monitor, and b) An ultrasound assisted designed brace and a smart brace device. Figure 1 shows the flow chart of the study. Each subject will have 50% chance of being in any one of the groups. An extra 15 minutes will be needed for both groups during the brace fitting clinic to install the brace monitor or smart brace device. An extra 30 minutes will be added to your casting. Participants will be monitored until the brace treatment is finished.

Detailed description: The brace monitor is a small electronic device which will be embedded inside the brace. It is a very low power system operating at 3.3 V and 2 milliampere (mA) (on average). It is able to store 12 months of data and the battery can last for 9 months. It will record how much time and how tightly the subject wears the brace. The brace with the monitor looks exactly the same as a standard brace. The subject won't feel any different and don't need to do anything beyond. We will replace the monitor with a new one at every standard follow up clinic.

A smart brace device is a small electronic device. It will have a small air bag embedded at the major pad area covered with stretchable leather. It will record how much time and how tightly the brace is worn. The air bag will inflate if the contact pressure between the brace and the body is lower than expected. The air bag will deflate if the contact pressure between the brace and the body is higher than expected. This automatic pressure adjustment will only be activated during daytime which is individualized based on the patient's sleep pattern. The system will also be activated only if breathing motion is detected (which means brace is worn). The smart brace monitor is able to store 6 months of data but requiring to recharge every day for 30 minutes. The smart brace monitor is a low power system (operating at 4.2 V and 150 mA max). It has an on-off switch and a pressure enable-disable regulation switch safety functions. Switching enable-disable regulation to off will make the smart brace device becomes a standard brace monitor. Turing off the on-off switch will disable all the functions and this brace will become a standard brace. We will replace the monitor with a new one at every standard follow up clinic.

The ultrasound assisted design requires to get 4 ultrasound images: normal standing, normal supine, bending left supine and bending right supine. Each scan takes approximately 1 minute. These 4 scans will provide spine flexibility information. After this, the subject will be asked to stand in a wooden positioning frame with pressure pads allow to move 3-dimensionally. Multiple adjustable brace pads will be applied to the patients' body according to orthotist suggestion. An ultrasound scan will be performed after the pads are applied. The orthotist will use the ultrasound image to decide if the pads are at the optimum locations and applied proper pressures. If the orthotist is satisfied with the correction, he/ she will use this setup to build the brace. Otherwise, he/she will adjust the position and orientation of the pads and repeated the ultrasound scan.

ELIGIBILITY:
Inclusion Criteria:

1. age 10 - 16 years
2. diagnosed of AIS
3. require full-time brace wear
4. have Cobb angle between 20° - 40°
5. have Risser sign ≤3
6. premenarchal or less than 1 year postmenarchal.

Exclusion Criteria:

1. patients who require surgery
2. presenting with associated musculoskeletal, neurological or other conditions possibly responsible for the curvature
3. physical or mental disability that prevent patients from complying with the bracing protocol

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2023-10 (Actual); Study Completion 2023-10 (Actual)

PRIMARY OUTCOMES:
Effectiveness of active brace treatment | 2 years after completing the brace treatment
  The proportions of successful treatment between two arms b to determine the overall effectiveness
Immediate Active effect | 1 year after enrollment
  Review the out of brace Cobb angle 1 year after using the spinal brace